CLINICAL TRIAL: NCT01415596
Title: The Effect of High Dose Salbutamol on Dynamic and Isometric Muscle Power and Recovery in Well-trained Males
Brief Title: The Effect of High Dose Salbutamol on Muscle Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Vibeke Backer, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: SALMUS2011
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-03

CONDITIONS: Ergogenic Effects of Salbutamol in Healthy Males
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Salbutamol (Active Comparator)
  Interventions: Drug: salbutamol

INTERVENTIONS:
Drug: salbutamol
  Arms: Salbutamol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Many athletes use beta2-agonists as treatment of airway hyperresponsiveness during exercise. High dose beta2-agonists may have an ergogenic effect on exercise performance. We hypotheis that the beta2-agonist, salbutamol, taken in high doses can improve muscle power and recovery during exercise in well-trained athletes.

ELIGIBILITY:
Inclusion Criteria:

* Males
* age 18-45
* training frequency > 10 hrs/wk
* informed consent

Exclusion Criteria:

* smoker or former smoker
* chronic diseases, as well as asthma
* allergy to the study drugs
* intake of any form of medicin or inhibited drugs during the study
* use of beta2-agonist 14 days before the intervention

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Muscle power

SECONDARY OUTCOMES:
Muscle recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen Northwest, Denmark